CLINICAL TRIAL: NCT00485498
Title: Managing Acute Schizophrenia, a Double Blind Comparison Between Two Atypical Antipsychotics - Olanzapine and Risperidone
Brief Title: Managing Acute Schizophrenia, a Comparison Between Two Atypical Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6704; F1D-GH-S036
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — olanzapine-fluoxetine combination; Risperidone

INTERVENTIONS:
Drug: Olanzapine Hydrochloride
Drug: Risperidone

SUMMARY:
The purpose of this study is to examine whether olanzapine, compared to risperidone, can provide more adequate and timely control of behavioral agitation in acutely ill subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 - 60
* Subjects must meet a clinical diagnosis of schizophrenia, schizophreniform disorder, or schizoaffective disorder according to DSM-IV
* Subjects' illness must not, in the opinion of the investigator, be caused by substance abuse
* BPRS total score (1 to 7 scale) of greater than or equal to 36 at visit 1
* Subjects must have a minimum total score of greater than or equal to 14 on the five items of the PANSS-EC and at least one individual item score of greater than or equal to 4 using the 1-7 scoring system prior to first dose of double-blind medications

Exclusion Criteria:

* Treatment with antipsychotics or benzodiazepines within 4 hours prior to the first study drug administration
* Treatment with an injectable depot neuroleptic within 1 injection interval prior to study drug administration
* Electroconvulsive therapy (ECT) within 1 month (90 days) prior to study entry (visit 1)
* Treatment with remoxipride within 6 months (180 days) prior to visit 1
* Documented history of allergic reaction to study medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2003-04; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
To determine if the efficacy of oral dose of olanzapine is greater than oral dose of risperidone in acute schizophrenia by comparing changes in agitation from baseline to 3 days post-first oral dose

SECONDARY OUTCOMES:
To assess the efficacy of olanzapine compared with risperidone, in reduction of scores from baseline to 3 days as measured by the BPRS-T, PANSS-P, ACES, CGI-I and CGI-S.
To assess the efficacy of olanzapine compared with risperidone, in reduction of scores from baseline to 6 weeks of acute treatment in the BPRS-T
To assess the efficacy of olanzapine compared with risperidone, in reduction of scores from baseline to 6 weeks of acute treatment in the PANSS
To compare the change in severity of akathasia in schizophrenic patients between olanzapine and risperidone as measured by the BAS within the 6-week treatment period
To compare the change of severity of extrapyramidal symptoms within the 6 week treatment with olanzapine and risperidone, as measured by the SAS

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing, China

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com